CLINICAL TRIAL: NCT04815902
Title: The Use of Senolytic and Anti-Fibrotic Agents to Improve the Beneficial Effect of Bone Marrow Stem Cells for Osteoarthritis
Brief Title: Use of Senolytic and Anti-Fibrotic Agents to Improve the Beneficial Effect of Bone Marrow Stem Cells for Osteoarthritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-15; 1UG3AR077748-01 (NIH)
Record Dates: First submitted 2021-03-17; First posted 2021-03-25 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Fisetin; Losartan; Osteoarthritis; Knee; Bone Marrow Concentrate; Bone Marrow Aspirate
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — fisetin; Losartan

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Fisetin and Active Losartan (Experimental): Losartan 12.5 mg, PO, BID beginning the first day after BMA Concentrate injection and continuing for 30 days. Fisetin 20mg/kg taken a total of 4 days prior to BMA Concentrate injection (-32 and -31 and -3 and -2) then again after BMA Concentrate injection a for a total of 6 days (32 & 33, 61 & 62 and 90 & 91).
  Interventions: Drug: Fisetin; Drug: Losartan
- Active Fisetin and Losartan Placebo (Active Comparator): Losartan Placebo 12.5 mg, PO, BID beginning the first day after BMA Concentrate injection and continuing for 30 days. Fisetin 20mg/kg taken a total of 4 days prior to BMA Concentrate injection (-32 and -31 and -3 and -2) then again after BMA Concentrate injection a for a total of 6 days (32 & 33, 61 & 62 and 90 & 91).
  Interventions: Drug: Fisetin; Drug: Placebo - Losartan
- Fisetin Placebo and Active Losartan (Active Comparator): Losartan 12.5 mg, PO, BID beginning the first day after BMA Concentrate injection and continuing for 30 days. Fisetin Placebo 20mg/kg taken a total of 4 days prior to BMA Concentrate injection (-32 and -31 and -3 and -2) then again after BMA Concentrate injection a for a total of 6 days (32 & 33, 61 & 62 and 90 & 91).
  Interventions: Drug: Losartan; Drug: Placebo Fisetin
- Control (Placebo Comparator): Losartan placebo 12.5 mg, PO, BID beginning the first day after BMA Concentrate injection and continuing for 30 days. Fisetin Placebo 20mg/kg taken a total of 4 days prior to BMA Concentrate injection (-32 and -31 and -3 and -2) then again after BMA Concentrate injection a for a total of 6 days (32 & 33, 61 & 62 and 90 & 91).
  Interventions: Drug: Placebo - Losartan; Drug: Placebo Fisetin

INTERVENTIONS:
Drug: Fisetin — Oral Fisetin 20 mg/kg taken for 10 days total.
  Other Names: Novusetin; 7,3',4'-flavon-3-ol; 3,3',4',7-tetrahydroxyflavone
  Arms: Active Fisetin and Active Losartan; Active Fisetin and Losartan Placebo
Drug: Losartan — 12.5 mg oral Losartan taken for 30 days total.
  Other Names: Losartan potassium
  Arms: Active Fisetin and Active Losartan; Fisetin Placebo and Active Losartan
Drug: Placebo - Losartan — Losartan appearance-matched microcrystalline cellulose placebo. 12.5 taken for 30 days total.
  Other Names: Placebo Oral Capsule
  Arms: Active Fisetin and Losartan Placebo; Control
Drug: Placebo Fisetin — Fisetin appearance-matched microcrystalline cellulose placebo. 20 mg/kg taken for 10 days total.
  Other Names: Placebo Oral Capsule
  Arms: Control; Fisetin Placebo and Active Losartan

SUMMARY:
This is a prospective, randomized, double-blind, active control clinical trial to evaluate the safety and efficacy of a senolytic agent (Fisetin) and an anti-fibrotic agent (Losartan), used independently and in combination, to improve beneficial effect demonstrated by the active control which is to be injection of autologous bone marrow aspirate concentrate (BMAC) into an osteoarthritic knee.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, active control clinical trial to evaluate the safety and efficacy of a senolytic agent (Fisetin) and an anti-fibrotic agent (Losartan), used independently and in combination, to improve beneficial effect demonstrated by the active control which is to be injection of autologous bone marrow aspirate concentrate (BMAC) into an osteoarthritic knee. 100 subjects with symptomatic unilateral or bilateral knee osteoarthritis (Kellgren-Lawrence grade II-IV) will be randomized into one of four arms (1:1:1:1). All subjects will receive an injection of BMAC. Group 1-n=25: Control (BMA concentrate + Fisetin Placebo + Losartan Placebo) Group 2-n=25: BMA concentrate + Fisetin Placebo + Active Losartan Group 3-n=25: BMA concentrate + Active Fisetin + Losartan Placebo Group 4-n=25: BMA concentrate + Active Fisetin + Active Losartan

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to personally give informed consent (consent via legally authorized representative will not be accepted) and who are willing to comply with all study-related procedures and assessments;
2. Between 40 and 85 years of age;
3. Ambulatory persons with osteoarthritis (OA) of at least one knee (Kellgren-Lawrence grade II-IV);
4. Baseline pain of 3-10 points on the target knee and a pain differential of at least -2 points on the contralateral knee as exhibited by the worst pain score (on the 11-point Numeric Rating Scale) for the previous week.

Exclusion Criteria:

Previous or Planned Knee Surgeries, Procedures and/or Treatments:

1. Planned surgery on either the contralateral or target knee at any time during the Study period including dosing and follow-up;
2. Within 6 months of signing informed consent has received diagnostic arthroscopy of the target knee or arthroscopic surgery (including microfracture and meniscectomy) on the target knee;
3. Within 12 weeks of signing informed consent has received intra-articular treatment of the target knee with steroids or hyaluronic acid derivatives;
4. History of previous total or partial arthroplasty in the target knee. Partial or total arthroplasty in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic;

   Current and/or Previous Medical Conditions, Surgeries and/or Procedures:
5. Within 2 years of signing informed consent history of active blood disorders (i.e., DVTs, chronic blood clotting, hemophilia, leukemia, myeloma, etc.); or active malignancy of any type or history of a malignancy (with the exception of subjects with a history of treated basal or squamous cell carcinoma);
6. Current diagnosis of fibromyalgia based on ACR criteria;
7. History of diabetes mellitus according to the American Diabetes Association criteria, or subjects previously diagnosed by a qualified physician as having diabetes (American Diabetes Association Standards of Medical Care in Diabetes 2016);
8. Any active known or suspected systemic autoimmune disease (except for vitiligo, residual auto-immune hypothyroidism requiring hormone replacement only, psoriasis not requiring systemic treatment for two years, conditions not expected to recur in the absence of an external trigger) or any history of a systemic inflammatory arthritis such as psoriatic, rheumatoid, ankylosing spondylitis or reactive arthritis;
9. Within 6 months of signing informed consent has undergone regenerative knee joint procedures including, but not limited to, platelet-rich plasma injections, mesenchymal stem cell transplantation, autologous chondrocyte transplantation, or mosaicplasty;
10. Current or prior history of other joint diseases including but not limited to joint dysplasia, crystal-induced arthropathy (such as gout, or calcium pyrophosphate deposition disease evidenced by clinical and/or radiographic means), aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler syndrome, joint infection, hemochromatosis, or neuropathic arthropathy of any cause;
11. Any medical condition, including findings in laboratory or medical history or in the baseline assessments, that (in the opinion of the Principal Investigator or his designee), constitutes a risk or contraindication for participation in the Study or that could interfere with the Study conduct, endpoint evaluation or prevent the subject from fully participating in all aspects of the Study;
12. Females who nursing a child, are pregnant or planning to become pregnant during study drug dosing;
13. Males who do not wish to abstain from sex with women of childbearing potential without use of contraceptive protection by either party during study drug dosing;
14. Unable to safely undergo an MRI based on MRI safety screening (for example, due to incompatible device/implant, severe claustrophobia, BMI greater than 40 kg/m2, or size exceeding the limits of the of the MRI equipment (coil and gantry);

    Current and/or Previous Medications and Supplements:
15. Taking medications that affect insulin activity, including Metformin or Acarbose within 1 week of signing informed consent;
16. Currently taking Losartan or Fisetin, allergy to any active or inactive ingredient of Losartan or Fisetin, and/or currently taking medication with known Losartan or Fisetin interaction;
17. Within 3 months of signing informed consent have taken senolytic agents including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
18. Subjects with any of the following drug/medication statuses:

    1. Currently taking Losartan;
    2. Currently taking Warfarin or related anticoagulants;
    3. Currently taking Lithium;
    4. Opioid analgesics taken in the past 8 weeks and are not willing to discontinue these medications through the duration of the study;
    5. Senolytic agents taken within the past 3 months and are not willing to discontinue these medications through the duration of the study, including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
    6. Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs;
    7. Subjects taking the following other drugs if they cannot be held (per the Principal Investigator) for at least 2 days before and during administration of Fisetin:

    cyclosporine, tacrolimus, repaglinide, and bosentan.
19. Taking a glucocorticoid within 1 month of signing informed consent;
20. Within 8 weeks of signing informed consent has used opioid analgesics, and are not willing to discontinue these medications through the duration of the study;
21. Within the 3 months of signing informed consent has received anticonvulsant therapy, pharmacological doses of thyroid hormone (causing decline of thyroid stimulating hormone below normal), calcium supplementation of > 1200 mg/d;
22. Within the 12 months prior to signing informed consent received any medications that affect bone turnover, including: adrenocorticosteroids (> 3 months at any time or > 10 days, estrogen (E) therapy or treatment with a selective E receptor modulator, or teriparatide;
23. Inability to tolerate oral medication;
24. Inadequate amount of BMA collected to serve the needs of the patient, ProofPoint Biologics and/or of the SPRI laboratory.

Behavioral Modification - Participants will be educated about the risk of excessive caffeine usage. Participants will be encouraged to reduce use by 50% prior to and during the Fisetin dosing days. Due to drug-drug interaction, subjects may not clear the caffeine from their system properly/as usual.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Adverse events will be collected from the date of BMAC injection to 12 months after injection
  Occurrence of adverse events

SECONDARY OUTCOMES:
Morphological and Quantitative Magnetic Resonance Imaging (MRI) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection)
  Cartilage quality assessed by blinded radiologist using morphological MRI. Quantitative MRI using T2 mapping images with texture analysis used to assess water content and collagen organization within the cartilage and surrounding tissue
Evaluation of patient reported outcome (PRO) for quality of life | within 3 months of injection, 32 days post baseline, 14 days post injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection, 18 months post injection
  12-question Short-Form General Health Survey (SF-12) - Including Physical Component Summary (PCS) and Mental Component Summary (MCS).
Evaluation of patient reported outcome (PRO) for knee functions (WOMAC) | within 3 months of injection, 32 days post baseline, 14 days post injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection, 18 months post injection
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) (24 questions; rated none, mild, moderate, or severe. Higher WOMAC score represents higher disability)
Evaluation of patient reported outcome (PRO) for knee functions (Tegner) | within 3 months of injection, 32 days post baseline, 14 days post injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection, 18 months post injection
  Tegner Physical Activity Scale (1 question; scale of 0 to10; 0 representing a low activity level and 10 representing a high activity level)
Evaluation of patient reported outcome (PRO) for knee functions (IKDC) | within 3 months of injection, 32 days post baseline, 14 days post injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection, 18 months post injection
  International Knee Documentation Committee (IKDC) Form. (scores range from 0 points or lowest level of function, to 100 points or highest level of function)
Patient-Reported Outcome Questionnaires | Screening, weekly post 1st study drug dose (pre-injection), weekly post injection (for 4 months)
  Numerical Rating Scale (NRS) for knee pain (6 questions with a scale of 0 to 10; 0 representing no pain and 10 representing extreme pain)
Change in muscle strength of the study knee | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection
  Isokinetic Dynamometry
Change in physical function of the Study Knee (LEK) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection
  Lower Extremity Kinematics
Change in physical function of the Study Knee (Stair Test) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection]
  Stair Test
Change in physical function of the Study Knee (fast 40-meter walk) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection
  Fast 40-meter walk
Change in physical function of the Study Knee (TUG) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection
  Timed up-and-go test
Change in physical function of the Study Knee (6-minute walk test) | 32 days - 3 months prior to injection, 6 months post injection, 12 months post injection]
  6-minute walk test
Change in associate biomarkers as compared to placebo in peripheral blood plasma/serum | screening, 14 days post-injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection
  Immunoassays for Biomarker assessment from blood serum. Analytes will be measured via immunoassays. The following analytes will be measured and reported in pg/ml. IL-1b, IL-6, IL-15, IL-1a, IL-1Ra, IL-7, IL-8, MCP-1, TNF-a , RANTES, VEGF, IFN-g, GRO, IP10, Eotaxin, PDGF-AA, PDGFAB-BB, EGF, FLT3L, GDF15, GDF11, FGF21, IL-18, SOST, OC, FGF-23, PTH, Leptin, Insulin, TIMP1, TIMP2, TGF-b1, TGF-b2, MMP-1, MMP-2, MMP-9, MMP-10, HA, COMP, CS846, CRP.
Change in CTX-II as compared to placebo in urine | 32 days post baseline, 6 months post injection, 12 months post injection
  Immunoassays for CTX-II detection in urine reported as pg/ml
Change in levels of senescent PBMCS (total and specific PBMC subsets such as T-Cells) | screening, 14 days post-injection, 30 days post injection, 3 months post injection, 6 months post injection, 12 months post injection
  Flow Cytometry based detection and quantification of senescent PBMCs isolated from whole blood. Intensity of the fluorescent marker C12FDG will be measured. Cells positive for C12FDG will be quantified and designated as senescent.
Change in synovial fluid content | 32 days post baseline, 6 months post injection, 12 months post injection
  Synovial Fluid Analysis
Characterization of Bone Marrow Derived Aspirate Concentrate cell content prior to injection | 32 days post baseline
  BMAC Analysis
Characterization of Bone Marrow Derived plasma biomarkers prior to injection | 32 days post baseline
  BMAC Analysis
Change in time to conversion to alternative treatment | Subjects may receive alternative treatment at any point during the 18-month study, continued participation will be determined on an individual basis (The time to resort to alternative therapy from baseline will be recorded)
  Alternative procedure as indicated. The time to resort to alternative therapy from baseline will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Huard, PhD, Principal Investigator — Steadman Philippon Research Institute; Marc Philippon, MD, Principal Investigator — Steadman Philippon Research Institute; Scott L Tashman, PhD, Principal Investigator — Steadman Philippon Research Institute
Locations (1):
- The Steadman Clinic, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No